CLINICAL TRIAL: NCT00871208
Title: Randomized, Placebo-Controlled Trial of Treatment of Atopic Dermatitis With Concurrent Altabax® and Topical Low-Potency Corticosteroids vs. Low-Potency Corticosteroid Mono-therapy
Brief Title: Trial of Treatment of Atopic Dermatitis With Concurrent Altabax® and Topical Low-Potency Corticosteroids Versus Low-Potency Corticosteroid Mono-therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLR08-057-111672
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; pruritus; quality of life
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — retapamulin; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Altabax (R) and Locoid Lipocream (R):Patients will apply both drugs sequentially to active lesions of atopic dermatitis. Physical examination, skin cultures, photos and quality of life scores will be performed at baseline, week 1, week 2 and week 4.
  Interventions: Drug: Altabax (R)
- 2 (Active Comparator): Vehicle and Locoid Lipocream (R):Patients will apply both drugs sequentially to active lesions of atopic dermatitis. Physical examination, skin cultures, photos and quality of life scores will be performed at baseline, week 1, week 2 and week 4.
  Interventions: Drug: Vehicle and Locoid lipocream (R)

INTERVENTIONS:
Drug: Altabax (R) — Retapamulin 1% ointment is to be applied to lesional atopic dermatitis twice-daily in addition to a topical corticosteroid (Locoid lipocream (R))
  Other Names: Altabax(R)ointment; Locoid lipocream (R)
  Arms: 1
Drug: Vehicle and Locoid lipocream (R) — The vehicle base of retapamulin ointment will be applied twice-daily to active lesions of atopic dermatitis in addition to locoid lipocream (R)
  Other Names: Locoid lipocream (R)
  Arms: 2

SUMMARY:
This study is designed to determine whether the addition of topical Altabax (R) to a treatment regimen of topical corticosteroid therapy speeds clearance of atopic dermatitis and improves quality of life.

DETAILED DESCRIPTION:
Background: Atopic dermatitis is a pruritic skin disorder which affects more than 10% of the United States population, one-third of whom report sleep disturbance and a quarter with chronic unremitting disease. Atopic dermatitis is a recurrent pruritic skin disorder which has a significant morbidity and extensive costs for the health care system. Quality of life is often impaired for patients with atopic dermatitis due to sleep disturbance, pruritus and the physical impairment of visible skin lesions.

The rapidity in which pruritus and lesional appearance are noted to resolve correlates strongly with improved patient satisfaction and improved quality of life.

Recently, a clinical trial of adding mupirocin into a regimen of topical corticosteroids has shown a significant enhancement in lesional clearance and symptom reduction with addition of mupirocin to the topical corticosteroid. These improvements were most notable within the first week of treatment.

Proposal: A 4-week clinical trial of 60 atopic dermatitis patients (ages 9 months to 17 years) would be conducted. All sixty patients would be given topical mid-potency corticosteroid (Locoid lipocream®) to be mixed with a second product. Half the patients would receive Altabax® and the other half would receive vehicle (blinded to subject and investigator). Patients would be advised to apply the topical randomized product first, let dry and then apply topical Locoid lipocream ® to affected areas, and then apply the topical randomized ointment product to each of the sites of skin disease on top of the Locoid lipocream ®. Treatment of affected areas would continue for 4 weeks or until lesions have cleared, which ever comes first. Parents of patients will be asked to maintain a written diary of drug application.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Atopic Dermatitis
2. Ages 9 months to 17 years
3. Presence of at least one lesion of atopic dermatitis at the time of baseline enrollment
4. Disease limited to less than 100 cm2 body surface area
5. EASI Score of at least 7, based on the Gong, et al publication Gong JQ, Lin L, Lin T, Hao F, Zeng FQ, Bi ZG, Yi D, Zhao B. Skin colonization by Staphylococcus aureus in patients with eczema and atopic dermatitis and relevant combined topical therapy: a double-blind multicentre randomized controlled trial. Br J Dermatol. 2006 Oct;155(4):680-7.

Exclusion Criteria:

1. Allergy to any ingredient in Altabax® or Locoid lipocream ®
2. Usage of oral corticosteroids within the 2 weeks prior to study initiation or during the study
3. Usage of topical corticosteroid or other topical prescriptions for atopic dermatitis in the week prior to study initiation
4. Inability to comply with the study protocol
5. Presence of major medical illness requiring systemic therapy including cancers.
6. Clinical diagnosis of bacterial infections of the skin, including impetigo or abscesses.

Ages: 9 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Superiority of drug to vehicle in reducing Eczema Area and Severity Index (EASI) scores in children with atopic dermatitis | Each patient will be enrolled for a 4 week trial

SECONDARY OUTCOMES:
Improved quality of life with usage of the drug altabax (R) and topical corticosteroids over vehicle and topical corticosteroids for treatment of atopic dermatitis in children with atopic dermatitis. | 4 week trial of medication

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Department of Dermatology, Beth Israel Medical Center, New York, New York
  - Department of Dermatology, Roosevelt Hospital, New York, New York
  - Department of Dermatology, St. Luke's-Roosevelt-Hospital Center, New York, New York

REFERENCES:
- [Background] Fivenson D, Arnold RJ, Kaniecki DJ, Cohen JL, Frech F, Finlay AY. The effect of atopic dermatitis on total burden of illness and quality of life on adults and children in a large managed care organization. J Manag Care Pharm. 2002 Sep-Oct;8(5):333-42. doi: 10.18553/jmcp.2002.8.5.333. PMID 14613399
- [Background] Carroll CL, Balkrishnan R, Feldman SR, Fleischer AB Jr, Manuel JC. The burden of atopic dermatitis: impact on the patient, family, and society. Pediatr Dermatol. 2005 May-Jun;22(3):192-9. doi: 10.1111/j.1525-1470.2005.22303.x. PMID 15916563
- [Background] Ricci G, Bendandi B, Bellini F, Patrizi A, Masi M. Atopic dermatitis: quality of life of young Italian children and their families and correlation with severity score. Pediatr Allergy Immunol. 2007 May;18(3):245-9. doi: 10.1111/j.1399-3038.2006.00502.x. PMID 17433002
- [Background] Gong JQ, Lin L, Lin T, Hao F, Zeng FQ, Bi ZG, Yi D, Zhao B. Skin colonization by Staphylococcus aureus in patients with eczema and atopic dermatitis and relevant combined topical therapy: a double-blind multicentre randomized controlled trial. Br J Dermatol. 2006 Oct;155(4):680-7. doi: 10.1111/j.1365-2133.2006.07410.x. PMID 16965415